CLINICAL TRIAL: NCT00528983
Title: A Phase 1, Open-label, Dose-Escalation Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Oral Azacitidine in Subjects With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML) or Acute Myelogenous Leukemia (AML).
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of Oral Azacitidine in Subjects With Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia and Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA PH US 2007 CL005
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes (MDS); Chronic Myelomonocytic Leukemia (CMML); Acute Myelogenous Leukemia (AML)
Keywords: Myelodysplastic Syndromes MDS; Acute Myelogenous Leukemia AML; Chronic Myelomonocytic Leukemia CMML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Juvenile | interventions — Injections, Subcutaneous; Azacitidine; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous (SC) Azacitidine and Oral Azacitidine (Experimental): Cycle 1 subjects receive SC Azacitidine for first 7 days of 28 day cycle. For Cycle 2 and beyond subjects receive Oral Azacitidine (experimental) for first 7 days of 28 day cycle.
  Interventions: Drug: Subcutaneous (SC) Azacitidine; Drug: Oral Azacitidine
- Oral Azacitidine (Experimental): Subjects receive Oral Azacitidine (experimental) QD or BID for the first 14 or 21 days of 28 day cycle.
  Interventions: Drug: Oral Azacitidine

INTERVENTIONS:
Drug: Subcutaneous (SC) Azacitidine — 75 mg/day for first 7 days of 28 day cycle for 1 cycle only.
  Other Names: Vidaza
  Arms: Subcutaneous (SC) Azacitidine and Oral Azacitidine
Drug: Oral Azacitidine — Cycle 2 and beyond starting dose of 120 mg/day for first 7 days of 28 day cycle. Dose will escalate in increments of 60 mg. Following evaluation dose escalation will occur in 120 mg increments until maximum tolerated dose (MTD) is reached.
  Other Names: CC-486
  Arms: Subcutaneous (SC) Azacitidine and Oral Azacitidine
Drug: Oral Azacitidine — Starting dose for 14 day-QD treatment schedule will be 300 mg/day. Starting dose for 14 day-BID, 21 day-QD, 21 day-BID treatment schedules will be 100 mg, 200mg, 300mg. Dose will escalate in increments of 100 mg until MTD is reached.
  Other Names: CC-486
  Arms: Oral Azacitidine

SUMMARY:
The purpose of this study is to determine whether a tablet form of azacitidine that taken by mouth is safe. This Phase I study will also look at different doses and different treatment schedules in order to better understand the effects (positive and negative) of oral azacitidine on the body and on the disease MDS, AML and CMML.

DETAILED DESCRIPTION:
Optional Extension Phase (OEP) to the AZA PH US 2007 CL 005 study which allows subjects who continue to receive oral azacitidine and have stable disease or are demonstrating clinical benefit as assessed by the Investigator, and have consented to participate, may enter the OEP of this study (at their current doses) at the start of their next cycle.

Subjects who are entering the OEP should be discontinued from Part 1 or Part 2 protocol prescribed therapy in the AZA PH US 2007 CL 005 study.

Subjects may continue to receive oral azacitidine in the OEP until they meet the criteria for study discontinuation or oral azacitidine becomes commercially available. Subjects discontinuing from the OEP will have an OEP discontinuation visit 28 days after the last dose of study drug or at study withdrawal.

Primary Objective of OEP is to evaluate long term safety of oral azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Diagnosis of low or Int-1 risk MDS
* Low platelet count, and/or low hemoglobin, and/or RBC transfusion-dependent and/or platelet transfusion-dependent
* ECOG Performance status 0-2
* Standard safety inclusion for serum creatinine, AST, ALT, bilirubin.
* Serum bicarbonate greater than or equal to 20 mEq/L.
* Use of acceptable birth control.
* Signed, written informed consent.

Exclusion Criteria:

* Diagnosis of acute PML.
* Previous or concurrent malignancy.
* Prior treatment with azacitidine or other demethylating agents.
* Treatment with any anticancer therapy or investigational drugs within 21 days.
* Hypersensitivity to azacitidine or mannitol.
* Presence of GI disease.
* Active, uncontrolled infection.
* Known Human Immunodeficiency Virus (HIV) or Hepatitis C, or known active viral Hepatitis B.
* Breastfeeding or Pregnant females;
* Presence of serious illness, medical condition, or other medical history which would be likely to interfere with a subject's participation in the study or with the interpretation of the results.
* Current congestive heart failure (NY Heart Association Class III-IV), unstable angina or angina requiring surgical or medical intervention within 6 months, myocardial infarct within 6 months, or uncontrolled cardiac arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-09-11 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2016-04-05 (Actual)

PRIMARY OUTCOMES:
Safety evaluation as measured by monitoring AEs, dose limiting toxicities, scheduled lab assessments, vital sign measurements, ECGs, & physical exams for study duration. Adverse changes in physical signs/symptoms will be graded according to CTC AE V.3.0. | 60 months
Maximum-tolerated dose | 60 months
Pharmacodynamic blood and bone marrow samples will be collected and evaluated. | 60 months

SECONDARY OUTCOMES:
Efficacy assessed by evidence of response (MDS subjects) and/or hematologic improvement (MDS subjects) examined using IWG criteria. | 60 months
Biologically active dose based on safety, PK and PD data. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Skikne, M.D., FACP; FCP (SA), Study Director — Celgene Corporation
Locations (18):
- United States (18):
  - University of Florida, Gainesville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Kansas University Medical Center, Westwood, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City VA Medical Center University of Kansas Medical Center, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology P.C., Albany, New York
  - Institute for Translational Oncology Research IRB, Greenville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Cancer Care, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - HOAST, San Antonio, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Yakima Valley Memorial Hospital/ North Star Lodge, Yakima, Washington

REFERENCES:
- [Background] Garcia-Manero G, Gore SD, Cogle C, Ward R, Shi T, Macbeth KJ, Laille E, Giordano H, Sakoian S, Jabbour E, Kantarjian H, Skikne B. Phase I study of oral azacitidine in myelodysplastic syndromes, chronic myelomonocytic leukemia, and acute myeloid leukemia. J Clin Oncol. 2011 Jun 20;29(18):2521-7. doi: 10.1200/JCO.2010.34.4226. Epub 2011 May 16. PMID 21576646
- [Background] Garcia-Manero G, Gore SD, Kambhampati S, Scott B, Tefferi A, Cogle CR, Edenfield WJ, Hetzer J, Kumar K, Laille E, Shi T, MacBeth KJ, Skikne B. Efficacy and safety of extended dosing schedules of CC-486 (oral azacitidine) in patients with lower-risk myelodysplastic syndromes. Leukemia. 2016 Apr;30(4):889-96. doi: 10.1038/leu.2015.265. Epub 2015 Oct 7. PMID 26442612
- [Derived] Laille E, Shi T, Garcia-Manero G, Cogle CR, Gore SD, Hetzer J, Kumar K, Skikne B, MacBeth KJ. Pharmacokinetics and Pharmacodynamics with Extended Dosing of CC-486 in Patients with Hematologic Malignancies. PLoS One. 2015 Aug 21;10(8):e0135520. doi: 10.1371/journal.pone.0135520. eCollection 2015. PMID 26296092